CLINICAL TRIAL: NCT02528006
Title: Treatment for Adductor Spasmodic Dysphonia by Type 2 Thyroplasty Using Titanium Bridges
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kumamoto University (Other)
Collaborators: Hokkaido University Hospital (Other); Yokohama City University Hospital (Unknown); Kyoto University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 001; otostl-0319 (Other: UMIN-CTR)
Record Dates: First submitted 2015-08-10; First posted 2015-08-19 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Adductor Spasmodic Dysphonia
Keywords: Spasmodic Dysphonia; Type 2 Thyroplasty; Titanium Bridges; Operation
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Titanium Bridges (Other): Surgery
  Interventions: Device: Type 2 Thyroplasty using Titanium Bridges

INTERVENTIONS:
Device: Type 2 Thyroplasty using Titanium Bridges

SUMMARY:
For adductor spasmodic dysphonia, there is a need for establishing a new therapy under the present circumstance where no standard therapy has been established yet and existing therapies fail to provide permanent effect. Evaluation of the efficacy of type 2 thyroplasty using titanium bridges will expand the therapeutic options available for adductor spasmodic dysphonia and establishment of a standard therapy.

DETAILED DESCRIPTION:
Spasmodic dysphonia is a type of functional dysphonia not associated with any organic abnormality or palsy of the larynx. The speech disorder in this disease is caused by involuntary and intermittent spasms of the intralaryngeal muscles (Castelon, 2002).

There is no curative treatment for this disease. Conservative therapies include voice training (voice therapy) and muscle relaxant medication to ease the tension in the larynx during speech, although there is not much evidence to support the effectiveness of either. An internationally employed therapy is local injection of botulinum toxin A into the intralaryngeal muscles to suppress involuntary movements of the vocal cords. The injection can be administered percutaneously from the anterior neck within a short time, and a number of reports have indicated a greater than 90% efficacy of this treatment (Tisch 2003, Blitzer 2010). However, this local injection therapy is effective only for a limited period of 3 to 4 months, and periodic injections have to be continued throughout life for maintaining relief from the symptoms under the present circumstances.

Type 2 thyroplasty is an operative procedure in which the thyroid cartilage is incised at the midline, and the incised gap is opened and fixed with the thyroarytenoid muscles attached on both sides, so that the vocal cords do not shut too tightly during speech even with strong adduction of the glottis, as the symptoms of adductor spasmodic dysphonia are caused by excessive closure of the glottis due to strong involuntary and intermittent adduction of the intralaryngeal muscles (Isshiki 2001).

In 2002, the titanium bridge made of biocompatible pure titanium was developed in Japan for exclusive use in type 2 thyroplasty (Isshiki 2004). When the titanium bridge was used in actual cases, the symptoms disappeared without recurrence after the operation (Sanuki 2007, Sanuki 2009, Isshiki & Sanuki 2009, Sanuki 2010).

There is a need for establishing a new therapy under the present circumstance where no standard therapy has been established yet and existing therapies fail to provide permanent effect. Evaluation of the efficacy of type 2 thyroplasty using titanium bridges will expand the therapeutic options available for adductor spasmodic dysphonia and establishment of a standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of adductor spasmodic dysphonia by a board certified otorhinolaryngologist certified by the Oto-Rhino-Laryngological Society of Japan, Inc.
2. At least 1 year experience of subjective or objective labored speech production, or pauses on certain sounds, due to adductor spasmodic dysphonia
3. A total score of 20 or more on the Voice Handicap Index-10 (VHI-10)
4. Non-responders to voice therapy performed before informed consent
5. 18 through 80 years of age inclusive at the time of informed consent
6. Written informed consent to participate in this study, provided by patients or their legally acceptable representatives

Exclusion Criteria:

1. Dysphagia, laryngeal paralysis, or any structural disorder in the vocal cord
2. Previous surgery for adductor spasmodic dysphonia
3. Local injection of botulinum toxin type A into the intralaryngeal muscles within 6 months before informed consent
4. Serious concomitant diseases
5. Surgery with general anesthesia scheduled during the study period or surgery performed within the past 4 weeks
6. Participation in any other study using any other intervention within 12 weeks before informed consent, or planned participation in such a study during the study period after enrollment in this study
7. Psychiatric disorder requiring treatment, or mental or intellectual disability that may affect the conduct of the study
8. A history of alcoholism or drug abuse
9. A history of hypersensitivity to pure titanium
10. Women who are pregnant or planning to become pregnant during the study period
11. Patients deemed ineligible for this study by the investigator for any other reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-07-27 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Change in VHI-10 scores assessed by Change from baseline in VHI-10 scores at 13 weeks after surgery | 13 weeks after surgery

SECONDARY OUTCOMES:
Changes in VHI,VHI-10 scores assessed by Changes in VHI-10 scores before and after surgery | 52 weeks after surgery
Changes in VHI,VHI-10 scores assessed by Changes in VHI scores before and after surgery | 52 weeks after surgery
Changes in VHI,VHI-10 scores assessed by Changes in VHI subscale scores in the functional (F), (P), and (E) | 52 weeks after surgery
Changes in VHI,VHI-10 scores assessed by Changes in phonatory function test results before and after surgery | 52 weeks after surgery
Changes in VHI,VHI-10 scores assessed by Changes in acoustic analysis results | 52 weeks after surgery
Changes in VHI,VHI-10 scores assessed by Frequency of adverse events and device defects | 52 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuji Sanuki, MD,PhD, Study Chair — Department of Otolaryngology,Kumamoto University
Locations (4):
- Japan (4):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Yokohama City University, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto

REFERENCES:
- [Background] Castelon Konkiewitz E, Trender-Gerhard I, Kamm C, Warner T, Ben-Shlomo Y, Gasser T, Conrad B, Ceballos-Baumann AO. Service-based survey of dystonia in munich. Neuroepidemiology. 2002 Jul-Aug;21(4):202-6. doi: 10.1159/000059525. PMID 12065883
- [Background] Ryuichi Yamazaki. Epidemiological Investigation on Spasmodic Dysphonia: Investigation by Questionnaire. The Japan Journal of Logopedics and Phoniatrics. 2001;42(4):343-347
- [Background] Sulica L. Contemporary management of spasmodic dysphonia. Curr Opin Otolaryngol Head Neck Surg. 2004 Dec;12(6):543-8. doi: 10.1097/01.moo.0000145959.50513.5e. PMID 15548915
- [Background] Ludlow CL, Adler CH, Berke GS, Bielamowicz SA, Blitzer A, Bressman SB, Hallett M, Jinnah HA, Juergens U, Martin SB, Perlmutter JS, Sapienza C, Singleton A, Tanner CM, Woodson GE. Research priorities in spasmodic dysphonia. Otolaryngol Head Neck Surg. 2008 Oct;139(4):495-505. doi: 10.1016/j.otohns.2008.05.624. PMID 18922334
- [Background] Tisch SH, Brake HM, Law M, Cole IE, Darveniza P. Spasmodic dysphonia: clinical features and effects of botulinum toxin therapy in 169 patients-an Australian experience. J Clin Neurosci. 2003 Jul;10(4):434-8. doi: 10.1016/s0967-5868(03)00020-1. PMID 12852881
- [Background] Blitzer A. Spasmodic dysphonia and botulinum toxin: experience from the largest treatment series. Eur J Neurol. 2010 Jul;17 Suppl 1:28-30. doi: 10.1111/j.1468-1331.2010.03047.x. PMID 20590805
- [Background] Schwartz SR, Cohen SM, Dailey SH, Rosenfeld RM, Deutsch ES, Gillespie MB, Granieri E, Hapner ER, Kimball CE, Krouse HJ, McMurray JS, Medina S, O'Brien K, Ouellette DR, Messinger-Rapport BJ, Stachler RJ, Strode S, Thompson DM, Stemple JC, Willging JP, Cowley T, McCoy S, Bernad PG, Patel MM. Clinical practice guideline: hoarseness (dysphonia). Otolaryngol Head Neck Surg. 2009 Sep;141(3 Suppl 2):S1-S31. doi: 10.1016/j.otohns.2009.06.744. PMID 19729111
- [Background] Tsuji DH, Chrispim FS, Imamura R, Sennes LU, Hachiya A. Impact in vocal quality in partial myectomy and neurectomy endoscopic of thyroarytenoid muscle in patients with adductor spasmodic dysphonia. Braz J Otorhinolaryngol. 2006 Mar-Apr;72(2):261-6. doi: 10.1016/s1808-8694(15)30066-5. PMID 16951863
- [Background] Nakamura K, Muta H, Watanabe Y, Mochizuki R, Yoshida T, Suzuki M. Surgical treatment for adductor spasmodic dysphonia--efficacy of bilateral thyroarytenoid myectomy under microlaryngoscopy. Acta Otolaryngol. 2008;128(12):1348-53. doi: 10.1080/00016480801965019. PMID 18607929
- [Background] Isshiki N, Haji T, Yamamoto Y, Mahieu HF. Thyroplasty for adductor spasmodic dysphonia: further experiences. Laryngoscope. 2001 Apr;111(4 Pt 1):615-21. doi: 10.1097/00005537-200104000-00011. PMID 11359129
- [Background] Isshiki N, Yamamoto I, Fukagai S. Type 2 thyroplasty for spasmodic dysphonia: fixation using a titanium bridge. Acta Otolaryngol. 2004 Apr;124(3):309-12. doi: 10.1080/00016480410016261. PMID 15141760
- [Background] Sanuki T, Isshiki N. Overall evaluation of effectiveness of type II thyroplasty for adductor spasmodic dysphonia. Laryngoscope. 2007 Dec;117(12):2255-9. doi: 10.1097/MLG.0b013e31814684fa. PMID 17921901
- [Background] Sanuki T, Isshiki N. Outcomes of type II thyroplasty for adductor spasmodic dysphonia: analysis of revision and unsatisfactory cases. Acta Otolaryngol. 2009 Nov;129(11):1287-93. doi: 10.3109/00016480802620639. PMID 19863326
- [Background] Isshiki N, Sanuki T. Surgical tips for type II thyroplasty for adductor spasmodic dysphonia: modified technique after reviewing unsatisfactory cases. Acta Otolaryngol. 2010 Feb;130(2):275-80. doi: 10.3109/00016480903036255. PMID 19513892
- [Background] Sanuki T, Yumoto E, Minoda R, Kodama N. Effects of type II thyroplasty on adductor spasmodic dysphonia. Otolaryngol Head Neck Surg. 2010 Apr;142(4):540-6. doi: 10.1016/j.otohns.2009.12.018. PMID 20304275
- [Background] Tetsuji Sanuki, Eiji Yumoto, Narihiro Kodama. Management of Adductor Spasmodic Dysphonia. The Larynx Japan. 2012;24(2):80-83
- [Background] Chan SW, Baxter M, Oates J, Yorston A. Long-term results of type II thyroplasty for adductor spasmodic dysphonia. Laryngoscope. 2004 Sep;114(9):1604-8. doi: 10.1097/00005537-200409000-00019. PMID 15475790
- [Background] Jacobson BH, Johnson A, Grywalski C, et al: The Voice Handicap Index (VHI): development and validation. Am J Speech-Lang Pathol, 1997; 6: 66-70.